CLINICAL TRIAL: NCT02329015
Title: Curriculum Evaluation of a Novel Health and Wellness Program Within New York City Schools
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Long Island University (Other)
Responsible Party: Principal Investigator, Marshall Hagins, Professor, Long Island University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SONIMA001
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Adolescent Behavior
Keywords: stress; alternative; complementary; self-regulation
MeSH Terms: conditions — Adolescent Behavior; Self-Control | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health and Wellness program (Experimental): Behavioral intervention
  Interventions: Behavioral: Yoga-informed Health and Wellness Program
- Physical Education Class (Active Comparator): Behavioral intervention
  Interventions: Behavioral: Physical Education Class

INTERVENTIONS:
Behavioral: Yoga-informed Health and Wellness Program — The HWP will be comprised of physical postures, breathing exercises, a period of sitting in stillness (meditation) and relaxation provided two times per week, 45 minutes per session, for the entire school year (Sept. - June).
  Arms: Health and Wellness program
Behavioral: Physical Education Class — Standard physical education
  Arms: Physical Education Class

SUMMARY:
The purpose of this study is to compare the academic and psycho-social benefits of a yoga-informed health and wellness program (HWP) to a standard physical education program for middle and high school students within New York City (NYC) schools.

DETAILED DESCRIPTION:
Approximately 100 students at a public New York City High School will be randomized at the level of class into either the experimental (yoga-informed health and wellness program) or control arm (physical education class). Students will receive two classes per week of approximately 45 minutes throughout the academic year. Data will be collected in September 2014 and February and May of 2015.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female students attending NYC schools

Exclusion Criteria:

* Lack of permission to attend physical education class

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Hagins, PhD, Principal Investigator — Long Island University
Locations (1):
- Eastside Community High School, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health and Wellness Program | Physical Education Class
Started | 48 | 64
Completed | 48 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health and Wellness Program | Physical Education Class | Total
Number analyzed (Participants) | 48 | 64 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (.94) | 15.4 (.98) | 15.3 (.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 19 | 39 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 7 | 5 | 12
  Black | 12 | 17 | 29
  Hispanic | 21 | 38 | 59
  White | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 48 | 64 | 112
Grade Point Average Previous Academic Year [Mean (Standard Deviation); unit: per cent] — GPA was calculated as the numeric average of course scores of all courses taken by the student weighted by credit load of each course using a standard process within NYC public schools
  per cent | 85.62 (7.9) | 83.38 (7.68) | 84.34 (7.81)
Height in inches [Mean (Standard Deviation); unit: inches] | 54.9 (5.7) | 57.5 (4.9) | 56.4 (5.23)
Weight [Mean (Standard Deviation); unit: pounds] | 129.5 (26.6) | 128.0 (21.9) | 128.64 (23.9)
Lunch Status [Number; unit: participants] — Data was not available for some participants relative to lunch status, therefore totals for each group do not equal baseline values
  participants
    Free lunch | 31 | 40 | 71
    Reduced Lunch | 6 | 11 | 17
    Full Price Lunch | 7 | 8 | 15
Cardiovascular Fitness (Pacer Test: Fitnessgram) [Mean (Standard Deviation); unit: Number of 20 meter laps completed] — The Pacer test is a test of aerobic fitness wherein participants are required to run back and forth on a level surface 20 meters in length. The allowed time to successfully complete each 20 meter run is gradually increased via an audible timer. The score represents the final number of runs successfully completed within the allowed time. Values range from 1-106 with higher values representing greater levels of aerobic fitness.
  Number of 20 meter laps completed | 48 (13.3) | 52.9 (17.3) | 50.8 (15.63)

OUTCOME MEASURES:

1. Primary Outcome: Academic Performance: Grade Point Averages
Description: GPA was calculated as the numeric average of course scores of all courses taken by the student weighted by credit load of each course using a standard process within NYC public schools.
Time Frame: 1 year
Population: Intent to treat analysis. Data from all participants was available at baseline and at end of study.
Measure: Mean (Standard Deviation); unit: per cent
Arm/Group | Health and Wellness Program | Physical Education Class
Number analyzed (Participants) | 48 | 64
per cent | 85.71 (8.44) | 83.45 (8.79)
Statistical Analysis 1: Comparison: Health and Wellness Program vs Physical Education Class; Model 1: An intent to treat analyses was performed determining effect of group assignment on academic performance while controlling for previous year GPA; Test type: Superiority or Other; p = 0.54, Regression, Logistic; Slope = 0.58, 95% CI 2-sided [-1.25 to 2.41]
Statistical Analysis 2: Comparison: Health and Wellness Program vs Physical Education Class; Model 2: As active participation between groups was significantly different a second intent to treat analysis was performed which added to Model 1 (controlling for previous year GPA) by controlling for active participation; Test type: Superiority or Other; p = 0.08, Regression, Linear; Slope = 1.67, 95% CI 2-sided [-0.21 to 3.55]
Statistical Analysis 3: Comparison: Health and Wellness Program vs Physical Education Class; Model 3: Per Protocol Analysis: it was hypothesized that any benefit of yoga education would only accrue if the student was assigned to yoga classes and actively participated in the class. A third Model was fit with an interaction term for class assignment and class participation; Test type: Superiority or Other; p = 0.009, Regression, Linear; Slope = 2.70, 95% CI 2-sided [0.69 to 4.71]

2. Secondary Outcome: Response to Stress Questionnaire (RSQ)
Description: A 57-item self-report questionnaire that was used as a measure of emotional regulation We examined two of the five constructs (24 of the 57 items) within the RSQ as these were most directly theoretically relevant to expected changes due to yoga practice: voluntary engagement and involuntary engagement. Higher values represent higher levels of negative stress responses. Values for the voluntary engagement subscale represent the mean value across 9 questions on the survey and values for the involuntary subscale represent the mean value across 15 questions on the survey. Values for each item range from 0-3, trherefore the total mean values reported as outcomes range from 0-3.
Time Frame: 1 year
Population: Missing data: 2 from experimental group, none from control group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health and Wellness Program | Physical Education Class
Number analyzed (Participants) | 46 | 64
units on a scale
  Involuntary Engagement | 0.84 (0.76) | 0.67 (0.64)
  Voluntary Engagement | 1.37 (0.61) | 1.27 (0.61)
Statistical Analysis 1: Comparison: Health and Wellness Program vs Physical Education Class; Analysis of the Voluntary subscale of the Response to Stress Questionnaire; Test type: Superiority or Other; p = 0.301, Regression, Linear

3. Secondary Outcome: Warwick Edinburgh Mental Well Being Scale
Description: A 14 item self-report measure assessing subjective well-being (1-5 scale). Higher values represent more positive mental well being. The summary measure is a sum of the 14 questions (not a mean). Summary values therefore range from 14-70.
Time Frame: 1 year
Population: 9 subjects missing from experimental group and 11 subjects missing from comparison group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health and Wellness Program | Physical Education Class
Number analyzed (Participants) | 39 | 53
units on a scale | 48.90 (13.44) | 49.51 (12.04)

4. Other Pre Specified Outcome: Self Report Questionnaire (Child and Adolescent Mindfulness Measure)
Description: A 10 item self-report measure assessing mindfulness skills (Scale 1-4). Items are reverse scored and summed (not mean). Higher scores mean more positive mindfulness skills. Min and maximum scores are 0-40.
Time Frame: 1 year
Population: 9 subjects missing from experimental group and 11 subjects missing from comparison group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health and Wellness Program | Physical Education Class
Number analyzed (Participants) | 39 | 53
units on a scale | 25.59 (8.72) | 26.38 (8.45)

5. Other Pre Specified Outcome: Student Self-Report Behavior Rating Inventory of Executive Function
Description: An 80 item self-report questionnaire assessing executive function and self regulation. The BRIEF-SR measures 8 non-overlapping clinical scales that measure different aspects of executive functioning with the Inhibit, Shift, Emotional control and Monitor subscales combining to create a Behavioral Regulation Index (BRI) and the Working Memory, Plan/Organize, Organization of Materials and Task Completion combining to create a Meta Cognition Index. These two indices combine to create a Global Executive Composite (GEC). Only the GEC was used within this study for analysis. Raw scores were converted to T scores (using gender and age for population norms) wherein a score of 50 represents the mean and a difference of 10 from the mean indicates a difference of one standard deviation.
Time Frame: 1 year
Population: 9 subjects missing from experimental group and 9 subjects missing from comparison group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health and Wellness Program | Physical Education Class
Number analyzed (Participants) | 39 | 55
units on a scale | 52.49 (13.84) | 46.84 (11.93)

6. Other Pre Specified Outcome: Teacher Report Behavior Rating Inventory of Executive Function
Description: Teacher reported 87 item questionnaire on students executive function and self regulation. The BRIEF for teachers measures 8 non-overlapping theoretically and empirically derived clinical scales that measure different aspects of executive functioning with the Inhibit, Shift, Emotional control and Monitor subscales combining to create a Behavioral Regulation Index (BRI) and the Working Memory, Plan/Organize, Organization of Materials and Task Completion combining to create a Meta Cognition Index. These two indices combine to create a Global Executive Composite (GEC). Only the GEC was used within this study for analysis Raw scores were converted to T scores (using gender and age for population norms) wherein a score of 50 represents the mean and a difference of 10 from the mean indicates a difference of one standard deviation.
Time Frame: One year
Population: 3 subjects missing from experimental group and 5 subjects missing from comparison group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health and Wellness Program | Physical Education Class
Number analyzed (Participants) | 45 | 59
units on a scale | 64.51 (20.40) | 59.39 (16.61)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Teachers were instructed to report to the PI any incident in which a student was injured during the intervention. Minor injuries not requiring a visit to the nurses station were not reported.
Arm/Group | Health and Wellness Program | Physical Education Class
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/64
Other Adverse Events (participants affected / at risk) | 0/48 | 0/64

LIMITATIONS AND CAVEATS:
This study had several limitations including the lack of blinding of tester and an excessive reliance on self-report. Analysis limited by an inability to test effects due to clustering. Novelty, Pygmalion, or motivational effect cannot be ruled out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No